CLINICAL TRIAL: NCT02441504
Title: Effects of Low Intensity Aerobic Exercise Training on the Microvascular Endothelial Function of Patients With Type 1 Diabetes: a Non-pharmacological Interventional Study
Brief Title: Effects of Low Intensity Aerobic Exercise on the Microvascular Endothelial Function of Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, ROGER DE MORAES, Dr. PhD, Instituto Nacional de Cardiologia de Laranjeiras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1988-CEP/HUPE
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Exercise training; microvascular rarefaction
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Microvascular Rarefaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low intensity exercise (Active Comparator): physical inactivity
  Interventions: Other: Low intensity Exercise

INTERVENTIONS:
Other: Low intensity Exercise — aerobic exercise training using walking and running

SUMMARY:
Background: The aim of the present study was to evaluate the changes in the microvascular density and reactivity in patients with type 1 diabetes (T1D) resulting from low intensity chronic exercise training.

Methods: This study included 22 (34 ± 7 years) consecutive outpatients with T1D and disease duration > six years. We used intravital video-microscopy to measure the basal skin capillary density as well as capillary recruitment using post-occlusive reactive hyperemia (PORH) in the dorsum of the fingers. Endothelium-dependent and -independent vasodilation of the skin microcirculation was evaluated in the forearm with a laser Doppler perfusion monitoring (LDPM) system in combination with acetylcholine and sodium nitroprusside iontophoresis, PORH and local thermal hyperemia.

DETAILED DESCRIPTION:
Subjects The present study was performed in accordance with the Helsinki Declaration of 1975, as revised in 2000, and the Institutional Review Board of the University Hospital of the State University of Rio de Janeiro, Brazil approved of this study. Once considered eligible, all subjects read and signed an informed consent document that was approved by the IRB.

Study subjects were recruited among patients who were followed up at a public hospital. Twenty-two individuals with T1D diagnosed for more than 6 years, between 25 and 50 years of age (mean 34 ± 7 years) were included in the study.

The initial clinical evaluation included the patient history and physical examination as well as recording of the following anthropometric data: weight, height, waist circumference and body mass index (BMI). Blood pressure measurements were collected with patients in the supine position after 5 minutes in quiet surroundings; they were repeated twice with two-minute intervals between measurements. All measurements were performed before and after twelve weeks of physical training.

Blood sampling and laboratory tests On the morning scheduled for the evaluation of cutaneous microcirculation, the patients presented in 12-hour fasted conditions for blood collection. Smokers should not have smoked or ingested caffeine from the night before until the completion of tests. The following variables were measured: fasting and postprandial plasma glucose, total cholesterol, LDL and HDL cholesterol, triglycerides, transaminases, high-sensitivity C-reactive protein, gamma-glutamyl transferase, creatine kinase, urea, creatinine, albumin and uric acid by colorimetric reactions with using a Cobas Mira-machine (Roche). Blood samples were collected before and after the physical training period. LDL cholesterol was calculated using Friedewald's formula. Serum samples were kept frozen at -80°C until measurement of the IL-6 levels with a commercial ELISA kit (Cayman Chemical Company, Ann Arbor, MI, USA), according to the manufacturer's instructions.

Physical training The study participants followed an aerobic training protocol targeted at low intensity and corresponding to 45% of the heart rate (HR) reserve [(HRmax - HRrest) x 45% + HRrest]. The exercise sessions were conducted 4 times per week for 12 weeks and included alternating walking and running, in accordance with the patient's fitness level, so that the heart rate reserve was between 40-50%. The heart rate was monitored using heart rate monitors (Polar Electro Oy, Kempele, Finland). In the first four weeks of training, there were additional increments of 10 minutes per session every week to promote gradual progression in the volume of 30 to 60 minutes during the remaining eight weeks.

Capillaroscopy by intra-vital videomicroscopy The capillary density, defined as the number of perfused capillaries per mm2 of skin area, was assessed by high-resolution intra-vital color microscopy (Moritex, Cambridge, UK) using a video microscopy system with an epi-illuminated fiber optic microscope containing a 100-W mercury vapor lamp light source and an M200 objective with a final magnification of 200X. The dorsum of the non-dominant middle phalanx was used for image acquisition, which occurred while the patient sat comfortably in a constant temperature environment (23±1°C). Images were acquired and saved for posterior off-line analysis using a semi-automatic integrated system (Microvision Instruments, Evry, France). The mean capillary density was calculated as the arithmetic mean of the number of visible (i.e., spontaneously perfused) capillaries in three contiguous microscopic fields of 1 mm2 each. A blood pressure cuff was then applied to the patient's arm and inflated to suprasystolic pressure (50 mm Hg above systolic arterial pressure) to completely interrupt blood flow for three minutes (post-occlusive reactive hyperemia test, PORH test). After cuff release, images were again acquired and recorded during the following 60-90 seconds, during which a maximal hyperemic response was expected to occur.

Microvascular reactivity to pharmacological stimulation The microvascular cutaneous reactivity was studied by laser Doppler perfusion monitoring (LDPM), a method that has previously been standardized and validated. Real-time variations in the cutaneous microcirculatory flow were assessed through an LDPM system (wavelength 780 nm; Periflux 5001, Perimed AB, Järfälla, Sweden) attached to a pharmacological micro-iontophoresis system (PeriIont, Perimed AB). The iontophoresis microelectrodes (PF 383, Perimed) were incorporated into the head of the laser probe (PF 481-1, Perimed), and the probe temperature was standardized to 32°C to avoid variations in the skin temperature and, consequently, in the measurements of microvascular flow. The drug-delivery electrodes were filled with 200 µl of 1% ACh solution (Sigma Chemical Co., USA) and placed on the ventral surface of the forearm, away from visible subcutaneous veins and areas of skin pigmentation. Neutral electrodes for current dispersion were placed 15 cm above the infusion electrodes, and reference points were marked and annotated to ensure reproducibility during the second examination, which took place at the end of the intervention period. After measuring the baseline flow for 5 minutes, four equal cumulative doses of ACh (anodal current) were applied at a constant intensity of 0.1 mA for 10, 20, 40 and 80 seconds, with total charges of 1, 2, 4 and 8 millicoulombs, respectively, allowing for a 120-second interval between doses. Recording of the microvascular flow induced by ACh was conducted for 10 minutes as follows: 2 minutes for each dose and 2 minutes to allow the flow to reach a plateau after the last dose. Using a new delivery electrode applied to a different location on the same forearm, four doses of a solution of 1% sodium nitroprusside (SNP; Sigma Chemical CO, USA) dissolved in distilled water were delivered using a cathodal current (same charges and intervals as for ACh).

The laser Doppler output, which is semiquantitative, is expressed in arbitrary perfusion units (PUs) of output voltage (1 PU = 10 mV) in accordance with general consensus (European Laser Doppler Users Groups, London, 1992). An area under the flow response to the ACh curve could be defined using the PeriSoft for Windows 2.5 software (Perimed, Järfälla, Sweden); this area was quantitatively measured and expressed in PU/s.

Microvascular reactivity to physiologic stimulation After measuring the resting capillary flow for 5 minutes using another laser probe (PF 457, Perimed) that had been positioned at the start of the recording session, the PORH test was performed. Following release of the pressure, the maximum flow and area under the PORH curve were measured. The mean value of the resting flow was considered the basal flow value. When the microvascular flow returned to the basal value after the PORH test (typically 5-10 minutes), the maximal skin microvascular vasodilatation was investigated with prolonged (20 minutes) local heating of the laser probe to 42°C. The baseline microvascular flux value was calculated as described above.

Statistical analysis The values were expressed as the means ± standard error of the means for the variables with a normal distribution and as median (percentiles 25th - 75th) for variables with a non-parametric distribution, according to results of the Shapiro-Wilk normality test. The data were analyzed by two-tailed paired t tests or the two-tailed Wilcoxon signed-rank test, as appropriate. The null hypothesis was rejected at P<0.05.

ELIGIBILITY:
Eligibility Gender: only male participants are being studied

Age Limits

Minimum 25 years

Maximum Age 50 years

Accepts Healthy Volunteers? no

Eligibility Criteria

Inclusion Criteria:

* Individuals with type 1 diabetes diagnosed for more than 6 years
* Age: between 25 and 50 years of age

Exclusion Criteria:

* Chronic renal disease

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Cutaneous Capillary Density in twelve weeks of aerobic physical activity | before and after 12 weeks of aerobic physical activity
  Chronic aerobic exercise has been involved in angiogenic processes that result in increased perfusion and capillary density. We believe that 12 weeks of aerobic exercise of low intensity is also able to exert the same effects in type 1diabetics patients. The microvascular cutaneous reactivity was studied by laser Doppler perfusion monitoring (LDPM), a method that has previously been standardized and validated. The capillary density, defined as the number of perfused capillaries per mm2 of skin area, was assessed by high-resolution intra-vital color microscopy using a video microscopy system with an epi-illuminated fiber optic microscope containing a 100-W mercury vapor lamp light source and an M200 objective with a final magnification of 200X.

REFERENCES:
- [Background] Matheus AS, Tibirica E, da Silva PB, de Fatima Bevilacqua da Matta M, Gomes MB. Uric acid levels are associated with microvascular endothelial dysfunction in patients with Type 1 diabetes. Diabet Med. 2011 Oct;28(10):1188-93. doi: 10.1111/j.1464-5491.2011.03349.x. PMID 21658123
- [Background] Gomes MB, Matheus AS, Tibirica E. Evaluation of microvascular endothelial function in patients with type 1 diabetes using laser-Doppler perfusion monitoring: which method to choose? Microvasc Res. 2008 Aug;76(2):132-3. doi: 10.1016/j.mvr.2008.04.003. Epub 2008 Apr 25. PMID 18533196
- [Background] Antonios TF, Nama V, Wang D, Manyonda IT. Microvascular remodelling in preeclampsia: quantifying capillary rarefaction accurately and independently predicts preeclampsia. Am J Hypertens. 2013 Sep;26(9):1162-9. doi: 10.1093/ajh/hpt087. Epub 2013 Jun 11. PMID 23757401
- [Background] Antonios TF, Kaski JC, Hasan KM, Brown SJ, Singer DR. Rarefaction of skin capillaries in patients with anginal chest pain and normal coronary arteriograms. Eur Heart J. 2001 Jul;22(13):1144-8. doi: 10.1053/euhj.2000.2442. PMID 11428855
- [Background] Nama V, Manyonda IT, Onwude J, Antonios TF. Structural capillary rarefaction and the onset of preeclampsia. Obstet Gynecol. 2012 May;119(5):967-74. doi: 10.1097/AOG.0b013e31824ea092. PMID 22525907
- [Derived] de Moraes R, Van Bavel D, Gomes MB, Tibirica E. Effects of non-supervised low intensity aerobic excise training on the microvascular endothelial function of patients with type 1 diabetes: a non-pharmacological interventional study. BMC Cardiovasc Disord. 2016 Jan 27;16:23. doi: 10.1186/s12872-016-0191-9. PMID 26817606